CLINICAL TRIAL: NCT03191123
Title: Resection Versus Transcatheter Arterial Chemoembolization for Hepatocellular Carcinoma With Solitary Huge Tumor: a Randomized Controlled Trial
Brief Title: Resection Versus Transcatheter Arterial Chemoembolization for Hepatocellular Carcinoma With Solitary Huge Tumor
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Huazhong University of Science and Technology (Other)
Responsible Party: Principal Investigator, Xiaoping Chen, Professor, Huazhong University of Science and Technology
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: chenxp008
Record Dates: First submitted 2017-06-14; First posted 2017-06-19 (Actual); Last update posted 2018-04-13 (Actual); Status verified 2018-04

CONDITIONS: Carcinoma, Hepatocellular; Survival Rate
Keywords: Hepatocellular Carcinoma; Hepatic Resection; TACE; Solitary Huge Tumor; Overall Survival
MeSH Terms: conditions — Carcinoma, Hepatocellular | interventions — Clinical Trials as Topic

STUDY DESIGN:
Who Masked: Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Hepatic resection (Active Comparator): Indications for Hepatic resection were the presence of appropriate residual liver volume determined by volumetric computed tomography and lack of hepatic encephalopathy.
  Interventions: Procedure: hepatic resection
- Transarterial Chemoembolization(TACE) (Experimental): Transarterial Chemoembolization is performed in less than one week after clinical diagnosis.
  Interventions: Procedure: TACE

INTERVENTIONS:
Procedure: hepatic resection — The aim of this intervention is to reach curative resection.
  Other Names: control
  Arms: Hepatic resection
Procedure: TACE — The aim of this intervention is one of the palliative treatment.
  Other Names: trial
  Arms: Transarterial Chemoembolization(TACE)

SUMMARY:
This clinical trial aims to compare hepatectomy with Transarterial Chemoembolization (TACE) for Hepatic Cellular Cancer With Solitary Huge Tumor (≥5cm). All patients will be divided into two group.One group will receive hepatic resection, while an another equivalent group patients will be treated with Transarterial Chemoembolization.

DETAILED DESCRIPTION:
Hepatocellular carcinoma (HCC) is the most common primary malignant tumor of the liver.For Barcelona Clinic Liver Cancer (BCLC) stage B patients，especially those with Solitary Huge Tumor (≥5cm) ，the better therapy between hepatic resection and transarterial chemoembolization remains controversial despite extensive studies。 From now on, we prospectively collected patients with solitary huge HCC who received hepatectomy or TACE. Of the 200 patients，100 patients were surgically treated and the others underwent TACE。After the treatment, patients received routine follow-up with physical examination, serum α-fetoprotein (AFP) level and ultrasonography at 3-month intervals for the first year and then every 6 months.The end of follow-up was determined as either the time of last follow-up (July 2019) or death. The overall survival，including 1, 2 and 3-year overall survival rates，will be analyse. All data are collected prospectively.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of Hepatic cellular Carcinoma.
* Patients with Solitary Huge Tumor (≥5cm）of Hepatic cellular Carcinoma (HCC) detected by Serum Alpha Fetoprotein (AFP) and CT or MRI.
* Patients without Hepatic vein or bile duct invasion and extrahepatic metastasis.
* Patients without surgical contraindication.
* Patients with Child A or B liver function and indocyanine green retention rate at 15min (ICGR15) < 10% before treatment.
* Laboratory examination: haemoglobin (Hb)>100g/L, white blood cell (WBC) > 3000/mL, blood platelet counts (PLT) > 8×10*10/L before treatment.
* Patients without severe esophagogastric varices before treatment.
* Patients with HBV，HBV DNA≤100, 000 copy/mL.
* All of the patients has written consent for this research.

Exclusion Criteria:

* Patients with multiple tumors or vascular or bile duct invasion or extrahepatic metastasis.
* Patients with surgical contraindication.
* Patients with Child C grade liver function before treatment.
* Patients with other malignancy.
* .Patients treated with hepatic resection or TACE before this treatment.
* Patients with severe esophagogastric varices or refractory ascites or coagulation dysfunction before treatment.

Ages: 20 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2016-07-05 (Actual); Primary Completion 2018-07-05 (Estimated); Study Completion 2019-07-05 (Estimated)

PRIMARY OUTCOMES:
3-year overall survival | 3 years
  Overall survival rate will be evaluated at 3 years after treatment

SECONDARY OUTCOMES:
1-year overall survival | 1 years
  Overall survival rate will be evaluated at 1 year after treatment
2-year overall survival | 2 years
  Overall survival rate will be evaluated at 2 years after treatment
Recurrence rates | 3 years
  any recurrence detected by CT, MRI and laboratory examination

OTHER OUTCOMES:
mortality | 30 days
  death within 30 days after surgery

CONTACTS AND LOCATIONS:
Locations (1):
- Hepatic surgery center, Tong ji Hospital, Wuhan, Hubei, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Yin L, Li H, Li AJ, Lau WY, Pan ZY, Lai EC, Wu MC, Zhou WP. Partial hepatectomy vs. transcatheter arterial chemoembolization for resectable multiple hepatocellular carcinoma beyond Milan Criteria: a RCT. J Hepatol. 2014 Jul;61(1):82-8. doi: 10.1016/j.jhep.2014.03.012. Epub 2014 Mar 17. PMID 24650695
- [Result] Metussin A, Patanwala I, Cross TJ. Partial hepatectomy vs. transcatheter arterial chemoembolization for resectable multiple hepatocellular carcinoma beyond Milan criteria: a RCT. J Hepatol. 2015 Mar;62(3):747-8. doi: 10.1016/j.jhep.2014.08.057. Epub 2014 Nov 7. No abstract available. PMID 25450210
- [Result] Jin YJ, Lee JW, Choi YJ, Chung HJ, Kim YS, Lee KY, Ahn SI, Shin WY, Cho SG, Jeon YS. Surgery versus transarterial chemoembolization for solitary large hepatocellular carcinoma of BCLC stage A. J Gastrointest Surg. 2014 Mar;18(3):555-61. doi: 10.1007/s11605-013-2440-x. Epub 2014 Jan 14. PMID 24420729